CLINICAL TRIAL: NCT01838629
Title: the Effect of Universal Salt Iodization on Thyroid Diseases
Status: Completed | Type: Observational
Sponsor: Weimin Xu (Other Government)
Responsible Party: Sponsor-Investigator, Weimin Xu, Superintendent of Department of Endemic Diseases Control and Prevention,Hangzhou Center for Disease Control and Prevention, Hangzhou, Zhejiang, China, Hangzhou Center of Disease Control and Prevention
Organization: Hangzhou Center of Disease Control and Prevention (Other Government)
Other Study IDs: 20090833B27
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The participants were invited to local community health center before 8:00 am after 8-hour fasting overnight. Firstly, each participant provided 10 ml spot urine samples. Then, 5 ml venous blood was collected using vacuum blood collection tube.

GROUPS / COHORTS (1):
- thyroid nodule

SUMMARY:
1. acquire the environmental iodine status of Hangzhou
2. acquire the iodine status of population in Hangzhou
3. acquire the prevalence of thyroid diseases in Hangzhou
4. explore the association between iodized salt and thyroid disease

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 6 years old;
2. living for above 5 years at present residence.

Exclusion Criteria:

1. resident with coronary angiography (CAG) or endoscopic retrograde cholangiopancreatography (ERCP) in 6 months;
2. resident taking amiodarone drug;
3. resident with abnormal kidney function or serious illness

Ages: 6 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted in Hangzhou, Zhejiang Province, China, which locates at east of China. This city covers eight districts and five counties. There are 8.7 millions residents in Hangzhou city; 73.25% of them living in urban areas, 26.75% in rural areas. This study was designed to be representative of the civilian from Hangzhou and collected information on demographic characteristics, health status, iodine intake and thyroid disease.
Sampling Method: Probability Sample
Enrollment: 12438 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
thyroid nodule | 8:00am (day 1)
  An ultrasound examination of the thyroid was performed to detect thyroid nodules, using a Sonoline Versa Pro (Siemens, Munich, Germany) with a 7.5-MHz, 70-mm linear transducer (effective length, 62 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Xu, Principal Investigator — Hangzhou Center for Disease Control and Prevention, Hangzhou, Zhejiang, China
Locations (1):
- Hangzhou Center of Disease Control and Prevention, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xu W, Chen Z, Li N, Liu H, Huo L, Huang Y, Jin X, Deng J, Zhu S, Zhang S, Yu Y. Relationship of anthropometric measurements to thyroid nodules in a Chinese population. BMJ Open. 2015 Dec 21;5(12):e008452. doi: 10.1136/bmjopen-2015-008452. PMID 26692553
- [Derived] Chen Z, Xu W, Huang Y, Jin X, Deng J, Zhu S, Liu H, Zhang S, Yu Y. Associations of noniodized salt and thyroid nodule among the Chinese population: a large cross-sectional study. Am J Clin Nutr. 2013 Sep;98(3):684-92. doi: 10.3945/ajcn.112.054353. Epub 2013 Jul 10. PMID 23842457